CLINICAL TRIAL: NCT02841592
Title: Non-rebreather at Flush Rate Compared to Bag Valve Mask With Assist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-preox_3
Record Dates: First submitted 2016-07-18; First posted 2016-07-22 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-rebreather (Active Comparator): This group will have a non-rebreather mask applied to the face and they will receive the flush rate oxygen intervention
  Interventions: Other: Flush rate oxygen
- Bag-valve-mask (Active Comparator): With each inspiration from the subject, the ventilation bag will be gently squeezed to provide positive pressure and augment the amount of oxygen that is received by the subject for each breath. This group will receive the flush rate oxygen with assist intervention.
  Interventions: Other: Flush rate oxygen with assist

INTERVENTIONS:
Other: Flush rate oxygen — Using a standard flowmeter (Precision Medical, 8MFA), the flow of oxygen will be fully opened and oxygen will be administered for three minutes.
  Arms: Non-rebreather
Other: Flush rate oxygen with assist — Using a standard flowmeter (Precision Medical, 8MFA), the flow of oxygen will be fully opened and oxygen will be administered for three minutes. Positive pressure breaths to match the subject's inspiration will be provided during the three minute period.
  Arms: Bag-valve-mask

SUMMARY:
This crossover investigation enrolls healthy volunteers and compares the exhaled oxygen content (FeO2) between the non-rebreather mask at the flush rate and a bag-valve-mask device at the flush rate, used with active positive pressure assistance.

ELIGIBILITY:
Inclusion Criteria:

* Age >17

Exclusion Criteria:

* Pregnant
* Any facial hair more than stubble that might impede a mask seal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Fraction of expired oxygen | 3 minutes
  The fraction of expired oxygen will be measured after three minutes of preoxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Driver BE, Klein LR, Carlson K, Harrington J, Reardon RF, Prekker ME. Preoxygenation With Flush Rate Oxygen: Comparing the Nonrebreather Mask With the Bag-Valve Mask. Ann Emerg Med. 2018 Mar;71(3):381-386. doi: 10.1016/j.annemergmed.2017.09.017. Epub 2017 Oct 28. PMID 29089172